CLINICAL TRIAL: NCT04407221
Title: COVID-19 Research in Organ Transplant Recipients
Acronym: CORONA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, John Søfteland, Consultant transplant surgeon, Vastra Gotaland Region
Other Study IDs: COV-19-SU-TX
Record Dates: First submitted 2020-05-03; First posted 2020-05-29 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Transplant Recipients
Keywords: Transplant Recipients; COVID-19 pandemic; COVID-19 virus; COVID-19 diagnostic testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Part 1:
  Plasma for serology PBMC
  Part 2:
  Plasma for serology PBMC Urine Stool NP or sputum swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is a global major public health emergency that disproportionately affects patients with risk factors such as advanced age, heart and lung disease, diabetes, hypertension, as well as compromised immunity. Despite the recent worldwide emergence of this disease and its rapid progression to a pandemic, very little is known about the risks facing solid organ recipients. The study aims to elucidate the prevalence of symptomatic, subclinical, and asymptomatic infection in the transplanted population by assessing their immunological response to SARS-CoV-2 infection. This will be studied seroepidemiologically in the whole cohort and retrospectively in transplanted patients admitted to hospital for COVID-19.

Primary objective: to elucidate the cumulative prevalence of SARS-CoV-2 infection in the transplanted population related to symptoms and hospitalizations; to assess the magnitude of immunological response and seroconversion kinetics for COVID-19. Secondary objectives: To examine the influence of medical parameters on COVID-19 infection and immune response such as: age, comorbidities current and recent pharmacological treatment, organ transplanted, and blood type, HLA genotype.

Study design:

Part 1: Longitudinal cohort study for seroepidemiology and disease burden. Part 2: Retrospective case-series for seroconversion kinetics and clinical course assessment.

Study population:

All solid organ transplanted patients in Sweden

DETAILED DESCRIPTION:
The study will assess the clinical course, the outcome, and the immunologic response of organ transplant patients who have had COVID-19 (participants); The investigators aim to study the development of the immune response to COVID-19 infection to see if participants on immunosuppressive treatment, will establish sufficient immunity to protect against reinfection. The findings among participants will be compared to a suitable control population. In addition, the investigators will identify patients in our cohort who are undergoing clinically apparent infections and study their clinical course and antibody response profile in the acute phase (seroconversion).

Control groups: Other current studies with matched protocols and WHO pooled data.

Overall study design Part 1: Potential participants are all patients who have undergone solid organ transplantation (SOT) in Sweden will be invited to participate in the longitudinal cohort seroprevalence part of the study (approximately 1000 patients will be included). This part of the study is a single-center longitudinal cohort study that will evaluate the development of antibodies against SARS-CoV-2 in solid organ recipients at all stages after transplantation and study their disease course, complications, and death rate.

The study has been designed to follow the best practices outlined by the WHO in their recent guidelines entitled "Population-based age-stratified seroepidemiological investigation protocol for COVID-19 virus infection COVID-19 v1.1". This will allow a comparison of symptoms, outcomes, case fatality rate, as well as antibody titers and prevalence, with other relevant control groups. Participant enrollment will be allowed for a maximum of 2 years. The duration of the study will be two years from enrollment. The last participant will thus complete follow-up a maximum of 4 years after the commencement of the study Part 2: The investigators will also do a retrospective assessment of transplanted patients in Sweden with PCR confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* A patient who has undergone solid organ transplantation in Sweden
* Must be able to take part in data reporting activities, sign the consent form, and submit blood samples at predefined intervals.

Exclusion Criteria:

-Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received a solid organ transplant can be offered to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 0 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 3 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 6 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 9 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 12 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 15 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 18 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 21 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Seroprevalence of SARS-Cov-2 antibodies (positive antibody test) | 24 months
  Cumulative presence of SARS-CoV-2 antibodies in plasma.
Change in levels of SARS-Cov-2 antibodies (antibody titers) | 0-24 months
  Change in titers of SARS-CoV-2 antibodies in plasma over time.

SECONDARY OUTCOMES:
Cellular response to SARS-Cov-2 (Th4 and Th8 levels) | 3 months
  PBMC specific responses, measured in PCR/serology positive patients.
Cellular response to SARS-Cov-2 (Th4 and Th8 levels) | 12 months
  PBMC specific responses, measured in PCR/serology positive patients.
Cellular response to SARS-Cov-2 (Th4 and Th8 levels) | 24 months
  PBMC specific responses, measured in PCR/serology positive patients.
Change in cellular response to SARS-Cov-2 (Th4 and Th8 levels) | 0-24 months
  Change in PBMC specific responses over time
Symptoms and hospitalisations (electronic questionnaire) | 0 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 3 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 6 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 9 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 12 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 15 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 18 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 21 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.
Symptoms and hospitalisations (electronic questionnaire) | 24 months
  Self-reported symptoms (WHO list of common COVID-19 symptoms) and hospitalisations during the past 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Oltean, MD, PhD, Study Chair — Transplant Institute, Sahlgrenska University; John M Søfteland, MD, PhD, Principal Investigator — Transplant Institute, Sahlgrenska University; Vanda Friman, MD, PhD, Study Director — Department of Infectious diseases, Gothenburg University
Locations (1):
- The Transplant Institute, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No